CLINICAL TRIAL: NCT01563367
Title: A Randomized, Prospective, Double-Blind, Comparative Placebo-Controlled Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by Infusions to Non-Anaemic Patients Undergoing Elective or Sub-Acute CABG, Valve Replacement or a Combination Thereof
Brief Title: A Prospective, Comparative Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by Infusions to Non-Anaemic Patients Undergoing Elective or Sub-Acute Coronary Artery Bypass Graft, Valve Replacement or a Combination Thereof
Acronym: CABG-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: CRO Max Neeman (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-Monofer-CABG-01
Record Dates: First submitted 2012-03-16; First posted 2012-03-27 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Non-anaemic Patients Undergoing Cardiac Surgery
Keywords: Anaemia; Cardiac surgery
MeSH Terms: conditions — Anemia | interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron isomaltoside 1000 (Monofer®) (Active Comparator): Iron isomaltoside 1000 (Monofer®) - Intravenous Infusion
  Interventions: Drug: Iron isomaltoside 1000 (Monofer®)
- 0,9% sodium saline (Placebo Comparator): Placebo (0.9% sodium saline) - Intravenous infusion
  Interventions: Drug: Natriumklorid 9 mg/ml, Fresenius Kabi

INTERVENTIONS:
Drug: Iron isomaltoside 1000 (Monofer®) — All subjects randomised to this group will receive 1000 mg iron isomaltoside 1000 as a single dose infusion administered over 15 minutes
  Arms: Iron isomaltoside 1000 (Monofer®)
Drug: Natriumklorid 9 mg/ml, Fresenius Kabi — All subjects randomised to this group will receive an infusion of 100 ml 0.9% sodium chlorid administered over 15 min.
  Other Names: 0.9% sodium chlorid.
  Arms: 0,9% sodium saline

SUMMARY:
The purpose of the study is to demonstrate that intravenous iron isomaltoside 1000 (Monofer®) is superior compared to placebo with respect to increasing the haemoglobin level in non-anaemic patients undergoing cardiac surgery

DETAILED DESCRIPTION:
The role of preoperative haemoglobin as a predictor of short-term and long-term outcomes after cardiac surgery has been well established. Anaemia can impede a patient's ability to recover fully and participate in postoperative rehabilitation. It has been found that patients with a normal haemoglobin level may become anaemic during surgery. An evaluation of patients undergoing cardiac surgery, i.e. CABG, valve or combined CABG-valve procedures showed that there was a decrease in mean haemoglobin level pre-surgery two and four days after surgery. To date, no prospective randomised clinical study in cardiac surgery assessing the effect of intravenous iron supplementation in patients undergoing cardiac surgery has been reported. This prospective, randomized, placebo controlled, double blind study is planned to evaluate the effect of intravenous iron isomaltoside 1000 (Monofer®) in comparison with placebo in non-anaemic patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Subjects undergoing elective or sub-acute CABG, valve replacement or a combination thereof
3. Female Hb ≥ 12.0 g/dl (7.45 mmol/l), Male Hb ≥ 13.0 g/dl (8.1 mmol/l).
4. Willingness to participate after informed consent.

Exclusion Criteria:

1. Subjects receiving blood transfusion less than 30 days before screening and/or during the elective or sub-acute CABG, valve replacement, or a combination thereof.
2. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
3. Serum Ferritin > 800 ng/ml.
4. Known hypersensitivity to any excipients in the investigational drug products.
5. Patients with a history of multiple allergies.
6. Decompensated liver cirrhosis and hepatitis.
7. Alanine Aminotransferase (ALT) > 3 times normal upper value.
8. Acute infections (assessed by clinical judgement).
9. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
10. Pregnant or nursing. (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: Contraceptive pills, Intrauterine Devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches).
11. Participation in any other clinical trial where the study drug has not passed five half-lives prior to screening.
12. Untreated Vitamin B12 or folate deficiency.
13. Other IV or oral iron treatment within 4 weeks prior to screening visit.
14. Erythropoietin treatment within 4 weeks prior to screening visit
15. Impaired renal function defined by se-creatinin > 150 µmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin (Hb) concentrations | From t=0 to t=4 weeks postoperatively
  To demonstrate that intravenous iron isomaltoside 1000 (Monofer®) is superior compared to placebo with respect to increasing the haemoglobin level in non- anaemic patients undergoing cardiac surgery

SECONDARY OUTCOMES:
Change in Hb concentrations | t=0, t=5 days and t=4 weeks
  Proportion of patients that are anaemic (women < 12 g/dL and men < 13 g/dL) at day 5 and week 4
Number of patients in each randomisation group who need blood transfusion and number of transfusions administered | From t=0 to t=day 5 and t=4 weeks
  To compare the number of patients who will need blood transfusion and number of transfusions in each randomisation group
Change in concentrations of serum ferritin, serum iron and Transferrin Saturation (TfS) TfS, and reticulocytes | Change from baseline (preoperatively- the day before surgery or same day) in concentrations of serum ferritin, serum iron and Transferrin Saturation (TfS) TfS, and reticulocytes at 4 weeks and 3 months postoperatively
  From t=0 to t=day 5 and t=4 weeks
Number of postoperative days to discharge | From t=0 to discharge
  To compare the number of days to discharge between the 2 randomisation groups
Changes in New York Heart Association (NYHA) classification | From t=0 to t=4 weeks
  To compare the changes in New York Heart Association (NYHA) classification from baseline to 4 weeks postoperatively
Number of patients in each randomisation group who experience any study drug related adverse events (AEs/SAEs/SUSARs) | From screening and until completion (t=-7 day and upto t=4 weeks)
  To compare the number of study drug related adverse events (AEs/SAEs/SUSARs) between subjects treated with iron isomaltoside 1000 (Monofer®) infusion and subjects treated with placebo infusion
Change in Hb | t=0, t=day 5 and t=week 4
  Proportion of patients able to maintain Hb between 9.5 and 12.5 g/dL (both values included) at day 5 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lykke Thomsen, Study Chair — Pharmacosmos A/S
Locations (1):
- Copenhagen, Denmark